CLINICAL TRIAL: NCT00395499
Title: Measurement of Risperidone and 9-Hydroxyrisperidone in Plasma and Saliva
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michael Aman, Professor Emeritus of Psychology, Ohio State University
Other Study IDs: 2000H0115
Record Dates: First submitted 2006-11-02; First posted 2006-11-03 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Patients Already Taking Risperidone for Clinical Indications
Keywords: Risperidone; 9-Hydroxyrisperidone; Plasma; Saliva; children
MeSH Terms: interventions — Risperidone

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: Risperidone

SUMMARY:
The purpose of this research is to: (1) examine the secrection of risperidone (RIS) (Risperdal) and its metabolite, 9-OH-RIS, in saliva, (2) determine the concentration ratio of RIS and 9-OH-RIS between plasma and saliva, and (3) compare the rate of decline in concentration of RIS and 9-OH-RIS in saliva and plasma by measurements at timed intervals during a single dosing interval.

DETAILED DESCRIPTION:
The purpose of this research is to: (1) examine the secrection of risperidone (RIS) (Risperdal) and its metabolite, 9-OH-RIS, in saliva, (2) determine the concentration ratio of RIS and 9-OH-RIS between plasma and saliva, and (3) compare the rate of decline in concentration of RIS and 9-OH-RIS in saliva and plasma by measurements at timed intervals during a single dosing interval.

RIS is a new atypical neuroleptic agent widely used in treatment of schizophrenia and related disorders. It is sometimes used in serious childhood disorders as well, such as autistic disorder. It has a beneficial effect on both positive and negative symptoms of schizophrenia, accompanied by a much lower incidence of adverse effects (e.g. parkinsonism, tardive dyskinesia, dystonias, neuroleptic malignant syndrome). RIS is also used as a treatment of children with pervasive developmental disorders (PDD). RIS is metabolized to 9-OH-RIS by hepatic CYP2D6 which exhibits genetic polymorphism. Since RIS and 9-OH-RIS are equally potent, the clinical significance of CYP 2D6 status is negligible. However, in extensive metabolizers (EM) the T(1/2) or RIS is about 3 hrs and taht of 9-OH-RIS is approximately 20 hrs. In poor metabolizers (PM) the half life of RIS is about 17 hrs and that of 9-OH-RIS 23 hrs.

Since compliance is a major problem in the management of schizophrenia, we are developing a rapid simplified test to measure RIS and 9-OH-RIS in salive and compare the concentration in samples of plasma collected concurrently. In this study, 12 adult patients (18 years and above) or minors (aged 5 to 17 years) already taking risperidone for clinical reasons will take their usual morning dose. Risperidone is usually administered once or twice a day.

At various intervals thereafter, a 1 to 2-milliliter specimen of saliva will be removed from the oral cavity by means of a syringe; in some cases it is more convenient to ask volunteers to expel saliva into a plastic cup. We will try to cover an 18-hour interval following dosing for the entire group (samples will be collected at 1/4, 1/2, 1, 2, 4, 8, 12, and 18 hours after taking the medicine. However, only some of the samples (2 or maximum of 3) will be gathered from any single patient. Following collection of saliva, a sample of 2 to 4 ml of blood will be withdrawn, and plasma will be separated and frozen. Saliva and plasma samples will gathered where the patient's drug concentrations would ordinarily be collected (e.g., Inpatient or Outpatient clinics, or phlebotomy laboratory). RIS concentrations will be measured by high pressure liquid chromatography (HPLC).

ELIGIBILITY:
Inclusion Criteria:

* aged 4 to 14 years, inclusive
* male or female
* any type of psychiatric diagnosis
* maintained on risperidone monotherapy for at least four weeks
* no medication adjustments for the last two weeks
* must be taking risperidone on a twice daily (morning and evening) schedule.

Exclusion Criteria:

* significant medical condition (e.g., heart disease, hypertension, liver or renal failure, pulmonary disease, unstable seizure disorder)
* females of child-bearing potential who score positive of pregnancy test
* receiving concurrent medications that may either bind to or are a substrate for CYP 450 2D6 or inhibit/induce CYP 3A3/4 activity. These include: anti-HIV medications, azole antifungal medications, calcium channel antagonists, carbamazepine, cimetidine, macrolide antibiotics (erythromycin, clarithromycin), phenytoin, propoxyphene, rifampin, or tramadol.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19
Dates: Start 2001-05; Study Completion 2003-04

CONTACTS AND LOCATIONS:
Overall Officials: Michael G. Aman, PhD, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - General Clinical Research Center, Columbus, Ohio
  - The Nisonger Center, Columbus, Ohio

REFERENCES:
- [Background] Aman MG, Paxton JW, Werry JS. Fluctuations in steady-state phenytoin concentrations as measured in saliva in children. Pediatr Pharmacol (New York). 1983;3(2):87-94. PMID 6674913
- [Background] Aman MG, Werry JS, Paxton JW, Turbott SH, Stewart AW. Effects of carbamazepine on psychomotor performance in children as a function of drug concentration, seizure type, and time of medication. Epilepsia. 1990 Jan-Feb;31(1):51-60. doi: 10.1111/j.1528-1157.1990.tb05360.x. PMID 2303013
- [Background] Aman MG, Werry JS, Paxton JW, Turbott SH. Effects of phenytoin on cognitive-motor performance in children as a function of drug concentration, seizure type, and time of medication. Epilepsia. 1994 Jan-Feb;35(1):172-80. doi: 10.1111/j.1528-1157.1994.tb02929.x. PMID 8112242
- [Background] Dumortier G, Lochu A, Zerrouk A, Van Nieuwenhuyse V, Colen de Melo P, Roche Rabreau D, Degrassat K. Whole saliva and plasma levels of clozapine and desmethylclozapine. J Clin Pharm Ther. 1998 Feb;23(1):35-40. doi: 10.1046/j.1365-2710.1998.00132.x. PMID 9756110
- [Background] Grant S, Fitton A. Risperidone. A review of its pharmacology and therapeutic potential in the treatment of schizophrenia. Drugs. 1994 Aug;48(2):253-73. doi: 10.2165/00003495-199448020-00009. PMID 7527327
- [Background] Haeckel R, Hanecke P. Application of saliva for drug monitoring. An in vivo model for transmembrane transport. Eur J Clin Chem Clin Biochem. 1996 Mar;34(3):171-91. PMID 8721405
- [Background] Lane HY, Chang WH. Risperidone-carbamazepine interactions: is cytochrome P450 3A involved? J Clin Psychiatry. 1998 Aug;59(8):430-1. No abstract available. PMID 9721825
- [Background] Lynn RK, Olsen GD, Leger RM, Gordon WP, Smith RG, Gerber N. The secretion of methadone and its major metabolite in the gastric juice of humans: comparison with blood and salivary concentrations. Drug Metab Dispos. 1976 Sep-Oct;4(5):504-9. PMID 10151
- [Background] Marder SR. Facilitating compliance with antipsychotic medication. J Clin Psychiatry. 1998;59 Suppl 3:21-5. PMID 9541334
- [Background] Nagasaki T, Ohkubo T, Sugawara K, Yasui N, Furukori H, Kaneko S. Determination of risperidone and 9-hydroxyrisperidone in human plasma by high-performance liquid chromatography: application to therapeutic drug monitoring in Japanese patients with schizophrenia. J Pharm Biomed Anal. 1999 Mar;19(3-4):595-601. doi: 10.1016/s0731-7085(98)00261-1. PMID 10704125
- [Background] Paxton JW, Aman MG, Werry JS. Fluctuations in salivary carbamazepine and carbamazepine-10,11-epoxide concentrations during the day in epileptic children. Epilepsia. 1983 Dec;24(6):716-24. doi: 10.1111/j.1528-1157.1983.tb04634.x. PMID 6641647
- [Background] Paxton JW, Donald RA. Enzyme immunoassay of carbamazepine in serum and saliva. J Pharmacol Methods. 1980 Jun;3(4):289-96. doi: 10.1016/0160-5402(80)90070-4. No abstract available. PMID 6993793
- [Background] Paxton JW, Whiting B, Stephen KW. Phenytoin concentrations in mixed, parotid and submandibular saliva and serum measured by radioimmunoassay. Br J Clin Pharmacol. 1977 Apr;4(2):185-91. doi: 10.1111/j.1365-2125.1977.tb00692.x. PMID 861132
- [Background] Walson PD, Mimaki T, Curless R, Mayersohn M, Perrier D. Once daily doses of phenobarbital in children. J Pediatr. 1980 Aug;97(2):303-5. doi: 10.1016/s0022-3476(80)80502-6. No abstract available. PMID 7400905
- [Background] Zuidema J, Hold KM, de Boer D, Maes RA. Saliva as a specimen for therapeutic drug monitoring in pharmacies. Pharm World Sci. 1996 Dec;18(6):193-4. doi: 10.1007/BF00735959. No abstract available. PMID 9010881